CLINICAL TRIAL: NCT01280253
Title: Can Biochemical Tests Predict Outcome in Patients With Hip Fracture?
Brief Title: Preoperative Biochemical Predictors of Outcome in Patients With Hip Fracture
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Anna and Edwin Berger Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: USILAN-2; 2010 (Other Grant/Funding Number: Anna och Edwin Berger Foundation); 1837 (Other Grant/Funding Number: Region Skane ALF)
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Hip Fracture
Keywords: Predictor; outcome; biochemical
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Litium-heparin plasma EDTA plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of the study is to identify biochemical predictors of morbidity and mortality in patients suffering from hip fracture. For this purpose blood samples are collected prehospitally or in the emergency department in patients with a suspected hip fracture. During the hospital stay medical history, anesthesiological management recorded. In addition, american society of anesthesiology physiological score (ASA), revised cardiac risk index (RCRI), and POSSUM score is calculated. Morbidity and mortality is recorded " in house", after 30 days, after 4 months and after 1 year. Biochemical predictors of outcome will be evaluated with logistic regression analysis. Biochemical predictors include pro-brain natriuretic peptide, lactate, pro-calcitonin, adrenomedullin, copeptin, cystatin c. The predictive value of the potential markers will be compared to that of ASA, RCRI and POSSUM.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with out of hospital hip fracture at University Hospital Lund Sweden
* Informed consent
* Blood sampling within 3 hrs of first contact with healthcare

Exclusion Criteria:

* No consent can be obtained
* Non-operative management
* Followup through the Swedish National Quality for Hip fracture patients not possible
* High energy trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting with hip fracture at University Hospital Lund Sweden
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days

SECONDARY OUTCOMES:
Morbidity | 30 day
  Infectious complications Cardiovascular complications Thromboembolic complications Respiratory complications Renal complications Surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skane University Hospital, Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request